CLINICAL TRIAL: NCT06455358
Title: 61Cu-NODAGA-LM3 PET/CT for the Detection of Neuroendocrine Tumors: The COPPER PET in NET Study A Prospective, Open-label, Randomized, Controlled, Single Centre, Phase I/II PET/CT Study
Brief Title: 61Cu-NODAGA-LM3 PET/CT for the Detection of Neuroendocrine Tumors (COPPER PET in NET)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2023-01981; th22Nicolas
Record Dates: First submitted 2024-05-30; First posted 2024-06-12 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-02

CONDITIONS: Neuroendocrine Tumors
Keywords: Radiolabeled somatostatin receptor ligands; SST PET/CT imaging; somatostatin receptor subtype 2 (SST2); Tumor detection
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — gallium Ga 68 dotatate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 61Cu-NODAGA-LM3 PET/CT before 68Ga-DOTATOC PET/CT (Experimental): Participants randomized into this group undergo 61Cu-NODAGA-LM3 PET/CT between 24 hours to 4 weeks before routine 68Ga-DOTATOC PET/CT.
  Interventions: Drug: 61Cu-NODAGA-LM3; Other: Comparator
- 61Cu-NODAGA-LM3 PET/CT after 68Ga-DOTATOC PET/CT (Experimental): Participants randomized into this group undergo 61Cu-NODAGA-LM3 PET/CT between 24 hours to 4 weeks after routine 68Ga-DOTATOC PET/CT.
  Interventions: Drug: 61Cu-NODAGA-LM3; Other: Comparator

INTERVENTIONS:
Drug: 61Cu-NODAGA-LM3 — Single intravenous administration of 61Cu-NODAGA-LM3 at an amount of 20 -40 μg (or 13 - 26 nmol) and an activity range of 150 MBq (±25%) followed by up to three PET/CT acquisitions.
Other: Comparator — Single intravenous administration of 68Ga-DOTA-TOC and PET/CT acquisitions as part of standard clinical care.
  Other Names: 68Ga-DOTA-TOC

SUMMARY:
The goal of this monocentric, open-label, randomized-controlled, reader-blind clinical study is to assess the safety of the radiolabeled somatostatin receptor ligand, 61Cu-NODAGA-LM3, and its sensitivity in comparison to the standard of care, 68Ga-DOTATOC, for PET/CT imaging in patients with well differentiated bronchopulmonary and gastroenteropancreatic neuroendocrine tumors.

DETAILED DESCRIPTION:
Neuroendocrine tumors (NET) originate from neuroendocrine cells and are most commonly found in the gastro-intestinal tract, pancreas and lung. Many NET grow slowly and are asymptomatic, leading to up to 50% being metastatic at diagnosis. Overexpression of somatostatin receptor subtype 2 (SST2) is a characteristic of NET and presents an important molecular target for the management of these tumors.

In Switzerland, two radiolabeled somatostatin analogues, gallium-68-labeled (68Ga)-DOTATOC and 68Ga-DOTATATE, are used for SST PET/CT imaging of well-differentiated neuroendocrine tumors. While these radiolabeled SST agonists provide high clinical performance and can be locally produced, they face limitations such as high costs, limited production capacity, short half-life hindering shipment to smaller centers, and high physiological uptake in organs like the liver, complicating tumor detection.

A novel copper-61 (61Cu) labeled somatostatin receptor antagonist, 61Cu-NODAGA-LM3, shows promise as an imaging agent for SST2 expressing tumors. It offers a longer half-life, enhanced tumor uptake and retention compared to established radiolabeled SST agonists, and improves image contrast.

This study aims to compare the safety and sensitivity of 61Cu-NODAGA-LM3 to the standard of care, 68Ga-DOTATOC, for SST PET/CT imaging in patients with well-differentiated bronchopulmonary and gastroenteropancreatic neuroendocrine tumors.

The results of the study potentially lead to enhanced diagnostic accuracy and patient care in the management of neuroendocrine tumors.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed
* >18 years old patients of either gender
* For women in child-bearing age: a negative pregnancy test is required
* Histologically proven well-differentiated bronchopulmonary (typical or atypical carcinoid) or gastroenteropancreatic neuroendocrine tumors (NET) of all grade (including NET G3 with Ki-67 <30 %)
* Clinical indication to somatostatin receptor (SST) PET/CT imaging for either primary staging, restaging, patient selection to Peptide Receptor Radionuclide Therapy, treatment planning or treatment response assessment
* Standard of care 68Ga-DOTATOC PET/CT performed or planned within max. 4 weeks prior or after IMP-administration, as clinically indicated
* At least 3 lesions detected by the previous somatostatin receptor scan, or if 68Ga-DOTATOC PET/CT is negative, a positive NETest not older than 4 weeks should be available in 5 additional patients
* Estimated eGFR (CKD-EPI) ≥ 45 mL/min
* If applicable, the last regular somatostatin analogue injection should be administered 2 weeks +/- 1 week prior to SST PET scan for long acting release forms

Exclusion Criteria:

* Known hypersensitivity to 61Cu, to NODAGA, to LM3 or to any of the excipients of 61Cu-NODAGA-LM3
* Prior or planned administration of a radiopharmaceutical within 8 half-lives of the radionuclide used on such radiopharmaceutical including at any time during the current study
* Initiation or continuation of active anti-tumor treatment between 61Cu-NODAGA-LM3 and 68Ga-DOTATOC PET/CT, except continuation of long acting somatostatin analogues
* Presence of active infection at screening or history of serious infection within the previous 6 weeks
* Pregnant or breast-feeding women
* History of somatic or psychiatric disease/condition that may interfere with the objectives and assessments of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events (number) | from Baseline up to 18 hours post injection
  The safety of 61Cu-NODAGA-LM3 is assessed in a primary safety analysis that is descriptive in nature and is performed in the safety analysis set, including information about the frequency (number) of adverse events.
Severity of adverse events assessed by CTCAE 5.0 | from Baseline up to 18 hours post injection
  The safety of 61Cu-NODAGA-LM3 is assessed in a primary safety analysis that is descriptive in nature and is performed in the safety analysis set, including information about the severity of adverse events.
  Severity will be graded as per CTCAE (Common Terminology Criteria for Adverse Events) Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting ageappropriate instrumental ADL (Activities of Daily Living).
  Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL.
  Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Assessment of the sensitivity of 61Cu-NODAGA-LM3 PET/CT | 1 hour post injection
  The sensitivity of 61Cu-NODAGA-LM3 PET/CT acquired ~ 1h p.i. is compared with that of the standard of care 68Ga-DOTA-TOC PET/CT acquired ~1h p.i..
  Sensitivity is determined based on the adjudication of all suspected lesions (union of the sets of lesions detected by two blinded independent readers) against a gold standard. The gold standard is defined either as a biopsy whenever possible and if clinically indicated or a comparison to the best imaging modality for the patient given case 2 - 7 months during follow up.
  After all "true" lesions are identified on all images, it is determined whether or not a given lesion has been identified on the 61Cu-NODAGA-LM3 PET/CT and on the 68Ga-DOTA-TOC PET/CT scans.

SECONDARY OUTCOMES:
Positive predictive value of 61Cu-NODAGA-LM3 PET/CT | 1 hour and 3 hours post injection
  The sensitivity of 61Cu-NODAGA-LM3 PET/CT acquired ~ 1h and ~ 3h p.i. is compared with that of the standard of care 68Ga-DOTA-TOC PET/CT acquired ~1h p.i. in the same patients.
  Sensitivity is determined based on the adjudication of all suspected lesions (union of the sets of lesions detected by two blinded independent readers) against a gold standard. The gold standard is defined either as a biopsy whenever possible and if clinically indicated or a comparison to the best imaging modality for the patient given case 2 - 7 months during follow up.
  After all "true" lesions are identified on all images, it is determined whether or not a given lesion has been identified on the 61Cu-NODAGA-LM3 PET/CT and on the 68Ga-DOTA-TOC PET/CT scans.
Dosimetry of 61Cu-NODAGA-LM3 | 1 hour, 3 and 18 hours post injection
  Whole body and healthy organ absorbed dose (Gy) is determined in 6 patients by acquiring 3 time-point PET/CT imaging (~1h, ~3 and ~18h p.i.)
Biodistribution of 61Cu-NODAGA-LM3 | 1 hour and 3 hours post injection
  Tracer uptake distribution in organs is assessed in 6 patients visually and quantitatively (organ SUVmax, SUVpeak and SUVmean) on 61Cu-NODAGA-LM3 PET/CT scans acquired at ~1h and ~3h p.i.
Peak plasma concentration (Cmax) of 61Cu-NODAGA-LM3 | Baseline, 2, 5, 10, 20, and 30 min, 1 hour, 2, 4, and 18 hours post injection
  The peak plasma concentration (Cmax) of 61Cu-NODAGA-LM3 is determined in 6 patients by serial blood sampling up to max. ~18 h.
Blood clearance of 61Cu-NODAGA-LM3 | Baseline, 2, 5, 10, 20, and 30 min, 1 hour, 2, 4, and 18 hours post injection
  The blood clearance of 61Cu-NODAGA-LM3 is determined in 6 patients by serial blood sampling up to max. ~18 h.
Area under the plasma concentration versus time curve (AUC) of 61Cu-NODAGA-LM3 | Baseline, 2, 5, 10, 20, and 30 min, 1 hour, 2, 4, and 18 hours post injection
  The area under the plasma concentration versus time curve (AUC) of 61Cu-NODAGA-LM3 is determined in 6 patients by serial blood sampling up to max. ~18 h.
Median of the median tumor uptake on 61Cu-NODAGA-LM3 PET/CT | 1 hour and 3 hours post injection
  The median of the mean tumor uptake (SUVmax) on 61Cu-NODAGA-LM3 PET/CT is determined at the best time-point for imaging and in comparison with 68Ga-DOTA-TOC PET/CT 1h p.i. for matched lesions only.
Median of the mean tumor to background ratio at the best time-point for imaging | 1 hour and 3 hours post injection
  The median of the tumor to background ratio on 61Cu-NODAGA-LM3 PET/CT at the best time-point for imaging is compared with 68Ga-DOTA-TOC PET/CT 1h p.i. for matched lesions only.
Differential Tumor detection rate | 1 hour and 3 hours post injection
  To determine the optimal imaging time-point, the difference between the tumor detection rate of 61Cu-NODAGA-LM3 PET/CT at ~1h and at ~3h p.i. is evaluated.
Mean tumor to background ratio | 1 hour and 3 hours post injection
  To determine the optimal imaging time-point, the mean of the tumor to background ratio of 61Cu-NODAGA-LM3 PET/CT performed ~1h and ~3h p.i. is compared for matched lesions only.
Mean signal to noise ratio | 1 hour and 3 hours post injection
  To determine the optimal imaging time-point, the mean signal to noise (SNR= SUVmax in Tumor VOI / Standard deviation in background VOI) of 61Cu-NODAGA-LM3 PET/CT is performed ~1h and ~3h post-injection for matched lesions only.
Interreader variability is assessed in terms of sensitivity; number of TP/(TP + FN) | 1 hour and 3 hours post injection
  To determine the optimal imaging time-point, the interreader variability is assessed in terms of sensitivity (sensitivity = number of true positive (TP) divided by the number of true positive and number of false negative (FN)) of 61Cu-NODAGA-LM3 PET/CT (1 vs 3 h p.i) and 68Ga-DOTATOC PET/CT is evaluated.
  Two independent blinded readers will assess the sensitivity of PET/CTs on a dedicated reading workstation using the software MIM Version 7.3.3.
Patient's preference | Baseline, 1 hour and 3 hours post injection
  To determine the optimal imaging time-point, the patient's preference is integrated by using a stress thermometer asking the patient to score their experience between the injection and scanning, and during scanning on a visual analogue scale, ranging from 0: not burdened at all to 10: extremely burdened.

OTHER OUTCOMES:
Optimal injected activity of 61Cu-NODAGA-LM3 | 1 hour and 3 hours post injection
  The optimal 61Cu-NODAGA-LM3 activity is determined by reconstructing the list-mode PET data for different acquisition frame duration. Signal-to-noise ratios are calculated for lung, pancreas, liver and small intestine as well as for at least one tumor lesion for matched lesions only.
Tumor detection rate of 61Cu-NODAGA-LM3 PET/CT | 1 hour and 3 hours post injection
  Tumor detection rate of 61Cu-NODAGA-LM3 PET/CT in 68Ga-DOTATOC PET/CT negative but NETest-positive NET patients is determined in max. 5 patients.
Correlation of tumor and organ uptake on 61Cu-NODAGA-LM3 PET/CT and quantitated post-treatment SPECT/CT | 1 hour and 3 hours post injection
  To correlate tumor and organ uptake visible on 61Cu-NODAGA-LM3 PET/CT and quantitated post-treatment SPECT/CT after targeted radionuclide therapy is attempted for 5 patients max.
Impact on management of 61Cu-NODAGA-LM3 PET/CT | 1 hour and 3 hours post injection
  To determine the impact on the clinical management of 61Cu-NODAGA-LM3 PET/CT in SST2-positive tumors, an analysis of pre-defined key imaging findings that may change the intended clinical management by tumor board decision is performed.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Nicolas, Dr., Principal Investigator — Division of Nuclear Medicine, University Hospital Basel
Locations (1):
- University Hospital Basel, Department of Radiology and Nuclear Medicine, Basel, Canton of Basel-City, Switzerland